CLINICAL TRIAL: NCT00351325
Title: A Phase I, Multiple Ascending Dose Study of BMS-663513, an Agonistic Anti-CD137 Monoclonal Antibody, Administered in Combination With Chemotherapy to Subjects With Advanced Solid Malignancies
Brief Title: A Study of BMS-663513 Administered in Combination With Chemotherapy to Subjects With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-004
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose escalation (Experimental)
  Interventions: Drug: BMS-663513

INTERVENTIONS:
Drug: BMS-663513 — mg/kg, IV, 0.3, 1, 3, 10 mg/kg, q 3 wks, up to 24 weeks

SUMMARY:
The purpose of this study is to assess the safety and tolerability of multiple escalating doses of BMS-663513 when given in combination with paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Good activity level
* Life expectancy of ≥ 6 months
* Solid tumor malignancy for which paclitaxel and carboplatin are appropriate

Exclusion Criteria:

* Major surgery within 4 weeks
* Any concurrent cancer
* History of autoimmune diseases
* Symptomatic bowel obstruction
* Continued use of steroids
* Symptomatic brain metastases
* Current nerve damage in fingers/toes
* Positive for HIV, hepatitis B/C
* White blood cells < 3,000
* Hemoglobin < 9
* Platelets < 100,000
* ALT/AST and/or alkaline phosphatase >= 2.5 x ULN
* Creatine > 1.5
* Prior BMS-663513

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending doses of BMS-663513 when given in combination with paclitaxel and carboplatin to subjects with advanced malignancies | throughout the study

SECONDARY OUTCOMES:
Explore PK and PD associations of BMS-663513 and the effect of BMS-663513 on immune system markers. | throughout the study
Describe anti-tumor activity | throughout the study
Obtain tissue or ascites for exploratory research | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (4):
  - University Of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital Of Upmc, Pittsburgh, Pennsylvania
  - University Of Virginia, Charlottesville, Virginia
  - University Of Washington, Seattle, Washington
- Local Institution, Toronto, Ontario, Canada